CLINICAL TRIAL: NCT00296023
Title: Low-Dose Allogeneic Peripheral Blood Stem Cell Transplantation for High-Risk Low Grade Hematologic Malignancies
Brief Title: Donor Stem Cell Transplant in Treating Older or Frail Patients With Hematologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000463724; UCSF-98251; UCSF-9805; UCSF-H9996-15837-06
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; noncontiguous stage II marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage II multiple myeloma; stage III multiple myeloma; chronic phase chronic myelogenous leukemia; primary myelofibrosis; polycythemia vera; prolymphocytic leukemia; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; chronic myelomonocytic leukemia; adult acute myeloid leukemia in remission; secondary acute myeloid leukemia; Waldenström macroglobulinemia; essential thrombocythemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; stage I multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Chronic-Phase; Primary Myelofibrosis; Polycythemia Vera; Leukemia, Prolymphocytic; Hodgkin Disease; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Waldenstrom Macroglobulinemia; Thrombocythemia, Essential; Congenital Abnormalities | interventions — Antilymphocyte Serum; Filgrastim; Busulfan; fludarabine phosphate; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell transplant (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: busulfan
Drug: fludarabine phosphate
Drug: methotrexate
Drug: tacrolimus
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and busulfan, before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and methotrexate and tacrolimus after the transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects of donor stem cell transplant in treating older or frail patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of non-myeloablative allogeneic peripheral blood stem cell transplantation, in terms of regimen-related organ toxicity and toxicity from acute graft-vs-host disease (GVHD), in older or medically frail patients with high-risk indolent hematologic malignancies.
* Determine overall survival, disease-free survival, and relapse risk at 1, 2, and 3 years post-transplantation in these patients.

Secondary

* Determine the engraftment of donor hematopoiesis at 6 weeks, 3 and 6 months, and 1 year post-transplantation in these patients.
* Determine the incidence and severity of chronic GVHD in older and medically infirm patients treated with this regimen.
* Determine the safety and efficacy of collecting peripheral blood stem cells from older donors (age > 60 years).
* Determine the need and efficacy of donor lymphocyte infusions in patients with residual disease after transplant.

OUTLINE:

* Non-myeloablative preparative regimen:Patients receive fludarabine IV over 30 minutes on days -7 to -3, busulfan IV over 2 hours every 8 hours on days -4 and -3, and anti-thymocyte globulin IV over 8 hours on days -4 to -1.
* Transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive tacrolimus orally every 12 hours or IV continuously beginning on day -2 and continuing until day 90, followed by a taper until day 180. Patients also receive methotrexate IV over 15-30 minutes on days 1, 3, 6, and 11.
* Donor lymphocyte infusions (DLIs): Patients with residual disease ≥ 6 months post-transplantation who are off immunosuppression for ≥ 30 days with no evidence of GVHD may receive DLIs. DLIs are administered ≥ 12 weeks apart in the presence of persistent disease, absence of severe (grade 3-4) GVHD, and absence of persistent GVHD after the first DLI.

After completion of study therapy, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a high-risk indolent hematologic malignancy meeting the following criteria:

  * Chronic lymphocytic leukemia (CLL) meeting 1 of the following criteria:

    * In second or subsequent remission
    * Failed to achieve a complete remission (CR) after chemotherapy
  * Non-Hodgkin's lymphoma (NHL) meeting 1 of the following criteria:

    * Low-grade NHL meeting 1 of the following criteria:

      * Standard-risk disease in second or subsequent remission
      * Standard-risk disease and failed to achieve a CR after chemotherapy
      * In first or subsequent remission with adverse International Prognostic Index (IPI) prognostic features, as defined by the presence of ≥ 3 of the following:

        * Age > 60 years
        * Tumor stage III or IV
        * Extranodal disease at > 1 site
        * ECOG performance status ≥ 2
        * Serum lactic dehydrogenase (LDH) > upper limit of normal (ULN)
    * Intermediate- or high-grade NHL meeting 1 of the following criteria:

      * In second or subsequent remission
      * Failed to achieve a CR after initial chemotherapy
  * Waldenstrom's macroglobulinemia meeting 1 of the following criteria:

    * In second or subsequent remission
    * Failed to achieve a CR after initial chemotherapy
  * Multiple myeloma meeting 1 of the following criteria:

    * In first or subsequent remission
    * Failed to achieve a CR after initial chemotherapy
  * Myeloproliferative disorders, including any of the following:

    * Chronic myelogenous leukemia in first or subsequent chronic phase
    * Myelofibrosis
    * Essential thrombocytopenia that is poorly responsive to standard therapy
    * Polycythemia vera that is poorly responsive to standard therapy or is in spent phase
  * Prolymphocytic leukemia meeting 1 of the following criteria:

    * In first or subsequent remission
    * Failed to achieve a CR after initial chemotherapy
  * Mantle cell lymphoma meeting 1 of the following criteria:

    * In first or subsequent remission
    * Failed to achieve a CR after initial chemotherapy
  * Hodgkin's lymphoma meeting the following criteria:

    * In second or subsequent remission

      * Prior remission duration > 6 months
    * No radiation therapy as the only prior primary therapy
  * Myelodysplastic syndromes (MDS) meeting 1 of the following criteria:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
    * Any MDS with transfusion dependence
    * Any MDS with ≥ 2 significant infections
  * Acute myeloid leukemia in morphologic remission
* In CR or partial remission or stabilization of disease after standard chemotherapy

  * No progressive or refractory disease
* Not eligible for standard allogeneic bone marrow transplantation
* Meets 1 of the following criteria:

  * Age 60 to 75 years old AND no co-morbid illness
  * Younger patients with any of the following comorbidities:

    * Decreased cardiac ejection fraction
    * Pulmonary dysfunction
    * Elevated liver function tests
    * Hepatitis C infection
    * Poor performance status
* Sibling or related donor available

  * Matched ≥ 5/6 HLA loci (A, B, and DR) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* ECOG performance status 0-2
* Creatinine < 2.0 mg/dL
* Creatinine clearance > 40 mL/min
* Ejection fraction > 30% by echocardiogram or MUGA
* Bilirubin < 3.0 mg/dL (if total bilirubin is elevated and Gilbert's disease is suspected, direct bilirubin must be normal)
* Alkaline phosphatase < 4 times ULN
* AST < 4 times ULN
* HIV negative
* Hepatitis B and/or C virus allowed if a liver biopsy (performed within the past 3 months) shows ≤ grade 2 inflammation
* No active infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-01; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Toxicity and survival | up to 36 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, MD, Principal Investigator — University of California, San Francisco; Willis Navarro, MD, Principal Investigator — University of California, San Francisco; Charles A. Linker, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - UCSF Comprehensive Cancer Center, San Francisco, California